CLINICAL TRIAL: NCT03020771
Title: Phase I Study to Evaluate Basic Pharmacodynamic, Pharmacological and Toxicological Effects of the Newly Developed Crimean-Congo Hemorrhagic Fever Vaccine for Humans, Prepared in Cell Culture and Inactivated With Formalin, and Administered Subcutaneously or Intramuscularly With Two Different Doses
Brief Title: Phase I Study to Evaluate Basic Pharmacodynamic, Pharmacological and Toxicological Effects of the Newly Developed Crimean-Congo Hemorrhagic Fever Vaccine for Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Scientific and Technological Research Council of Turkey (Other)
Collaborators: MonitorCRO (Industry)
Responsible Party: Principal Investigator, Aydin Erenmemisoglu, MD PhD, The Scientific and Technological Research Council of Turkey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MON116.40.1
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Crimean-Congo Hemorrhagic Fever
Keywords: Crimean-congo hemorrhagic fever; vaccine; human; phase I
MeSH Terms: conditions — Hemorrhagic Fever, Crimean

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 5 mcg IM (Active Comparator)
  Interventions: Biological: KIRIM-KONGO-VAX
- 5 mcg SC (Active Comparator)
  Interventions: Biological: KIRIM-KONGO-VAX
- 5 mcg IM control (Placebo Comparator): 0.9% NaCl Solution
  Interventions: Other: Placebo
- 5 mcg SC control (Placebo Comparator): 0.9% NaCl Solution
  Interventions: Other: Placebo
- 10 mcg IM (Active Comparator)
  Interventions: Biological: KIRIM-KONGO-VAX
- 10 mcg SC (Active Comparator)
  Interventions: Biological: KIRIM-KONGO-VAX

INTERVENTIONS:
Biological: KIRIM-KONGO-VAX — Crimean-Congo Hemorrhagic Fever Vaccine
  Arms: 10 mcg IM; 10 mcg SC; 5 mcg IM; 5 mcg SC
Other: Placebo
  Arms: 5 mcg IM control; 5 mcg SC control

SUMMARY:
This study covers the first trial of the Crimean-Congo Hemorrhagic fever virus (CKKA) vaccine on humans (healthy volunteers), which has been developed in Turkey and has completed preclinical toxicology studies to be performed on experimental animals. Also, this study is a Phase I, randomized, double-blind, national, single-center, placebo-controlled study that is designed to evaluate the safety and efficacy of the CKKA vaccine. A total of 60 (12 + 48) healthy male and/or female volunteers will be participating in this study, and the study is planned to last approximately one year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, white in the 18-55 age range, men and/or women who agree not to become pregnant until 2 months after the start of the last vaccination
* Body weights are at limits to exclude anorexia or obesity (The BMI limits accepted for this study are 18.5-30 kg /m2)
* According to clinical and standard laboratory tests, physical and spiritually healthy volunteers.

Exclusion Criteria:

* The 20 days before the study any vaccination applied volunteers
* Persons with clinically significant liver, kidney, gastrointestinal, cardiovascular, psychiatric, pulmonary, hematologic, endocrinological, or other significant acute or chronic abnormalities in the medical history of the volunteer or in the examination.
* Volunteers who have previously had any pulmonary infection or have previously used immunosuppressive drugs (including corticosteroids) for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety of the IMP in terms of number and frequency of any adverse events, any abnormal findings in physical examinations, ECGs, and laboratory parameters occurred during the follow up period. | One year follow up
  The safety parameters planned for this experimental vaccine will be all adverse events experienced by the volunteers or not identified by the volunteer and identified resulting from physical examinations or laboratory tests or ECG by the investigators.

SECONDARY OUTCOMES:
Immunogenicity | One year follow up
  This secondary outcome will be performed at every humoral and cellular level after each immunization, based on immunological responses.

CONTACTS AND LOCATIONS:
Overall Officials: Aydın Erenmemisoglu, MD PhD, Principal Investigator — TC Erciyes University